CLINICAL TRIAL: NCT02578446
Title: Migration and Survival of the Uncemented Tritanium Tibia Compared With the Cemented Metal-backed Tibia Using the Triathlon Cruciate Retaining (CR) Total Knee System. A Single Centre RSA Study
Brief Title: Uncemented Tritanium Compared With Cemented Metal-backed Tibia Components in Total Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Leiden University Medical Center (Other); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K-I-058
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Arthroplasty; Replacement; Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncemented Triathlon Tritanium CR (Experimental): Primary total knee replacement with Uncemented Triathlon Tritanium CR Total Knee System
  Interventions: Device: Uncemented Triathlon Tritanium CR Total Knee System
- Cemented Triathlon CR (Active Comparator): Primary total knee replacement with Cemented Triathlon CR Total Knee System
  Interventions: Device: Cemented Triathlon CR Total Knee System

INTERVENTIONS:
Device: Uncemented Triathlon Tritanium CR Total Knee System — Primary Total Knee Replacement
  Other Names: Stryker Orthopaedics
  Arms: Uncemented Triathlon Tritanium CR
Device: Cemented Triathlon CR Total Knee System — Primary Total Knee Replacement
  Other Names: Stryker Orthopaedics
  Arms: Cemented Triathlon CR

SUMMARY:
The optimal method of total knee replacement component fixation to the bone remains a challenge. The use of bone cement is considered the gold standard and is the preferred technique for most surgeons. However, uncemented fixation methods have been developed in an attempt to tackle problems that can be seen when cement is used. The cement-bone interlock can deform and degrade over the years and can lead to aseptic loosening, especially in young and active patients. A loosened prosthesis results in an impaired functioning and painful knee in daily life for which a revision of the prosthesis may be necessary. To prevent aseptic loosening and subsequent revision surgery, new methods of uncemented fixation have been developed.

One of these methods is to use a highly porous metal called Tritanium®. It can improve the biologic fixation by resembling the characteristics of trabecular bone. It is expected that this surface aids bone ingrowth and to have similar or even better results concerning early fixation properties and long-term durability compared with cemented fixation. Excellent results using this highly porous Tritanium have been seen in total hip surgery already.

This single-blinded, randomized clinical trial will assess clinical and radiological outcomes including Roentgen Stereophotogrammetry (RSA) measurements of a newly approved uncemented Triathlon Tritanium CR total knee prosthesis compared with a standard cemented Triathlon metal-backed CR total knee prosthesis (both by Stryker Orthopaedics). Two arms of each 35 patients will be included.

The primary outcome measure will be prosthetic migration after two years of the uncemented Triathlon Tritanium CR Total Knee and the cemented Triathlon CR Total Knee by means of RSA. It is hypothesized that the new uncemented Tritanium prosthesis will perform at least equally good in terms of migration and clinical parameters compared with the standard cemented Triathlon.

The secondary outcome measure will be long-term (10-year) survival based on the two-year migration patterns combined with clinical factors and radiographic aspects. In order to identify other clinical parameters besides the fixation of the prosthesis components, clinical scores and radiographic aspects will be correlated with the RSA outcome. The 10-year results will be used to verify the predicted long-term survival results.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to understand the meaning of the study and is willing to sign the Ethics Commission (EC) approved, study specific Informed Patient Consent Form.
2. Patients eligible and scheduled to undergo primary total knee replacement with any of the following indication.

   * Painful and disabled knee joint resulting from osteoarthritis (Ahlbäck stage II to V)
   * One or more compartments are involved.
3. Ability and willingness to follow instructions, including control of weight and activity level, and to return for follow-up evaluations.
4. A good nutritional state of the patient.
5. The subject is a male or non-pregnant female between 40 and 75 years of age.

Exclusion Criteria:

1. The subject is morbidly obese, defined as Body Mass Index (BMI) of > 37.
2. Previous major knee surgery
3. Patients who had a Total Knee Arthroplasty (TKA) on contralateral side within the last 6 months that is considered to have an unsatisfactory outcome. (Patients with contralateral TKA > 3 months ago with good outcome can be included in the study).
4. Patients with other severe concurrent joint involvements that can affect their outcome.
5. Patient has a flexion contracture of 15° and more.
6. Patient has a varus/valgus contracture of 15° and more.
7. The subject will be operated bilaterally.
8. The subject has an active or suspected latent infection in or about the knee joint.
9. Osteomyelitis
10. The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
11. The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
12. The subject is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
13. Female patients planning a pregnancy during the course of the study.
14. The patient is unable or unwilling to sign the Informed Consent specific to this study.

Secondary exclusion criteria: when there are less than five tibia-bone markers or less than three insert markers visible in the baseline RSA photograph and it will not improve by placing the patient in another position, the patient will be excluded from the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Migration, measured by means of RSA | 2 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)

SECONDARY OUTCOMES:
Migration, measured by means of RSA | 10 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)
Investigation of clinical performance and patient outcome with the Knee Society Score (KSS) | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Investigation of clinical performance and patient outcome with the Knee Injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Investigation of clinical performance and patient outcome with EuroQuol-5 dimension (EQ-5D) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
Investigation of clinical performance and patient outcome with the Forgotten Joint Score (FJS) patient questionnaire. | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The FJS consists of 12 questions and focuses on the patients' awareness of their joint replacement during a range of day to day and recreational activities. The score has a range of 0-100.questionnaire
Investigation of patient outcome with radiographic analysis | 3 months, 1, 2, 5, 7 and 10 years
  Plain radiographs will be obtained for assessment of fixation of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Sören Toksvig-Larsen, Ass Prof, Principal Investigator — Department of Orthopaedics Hässleholm-Kristianstad-Ystad, Hässleholm Hospital
Locations (2):
- Leiden University Medical Center, Leiden, Netherlands
- Department of Orthopaedics Hässleholm-Kristianstad-Ystad, Hässleholm Hospital, Hässleholm, Sweden